CLINICAL TRIAL: NCT06213155
Title: A Randomized, Parallel Arm, Sham-controlled, Double-blinded, Investigator-initiated Trial to Investigate the Safety and Efficacy of Percutaneous Peripheral Cryoneurolysis Therapy in Medically Refractory Trigeminal Neuralgia: a Pilot Study
Brief Title: A Study to Investigate the Efficacy of Pain Reduction With Cryoneurolysis Compared With Sham-treatment in Adults With Trigeminal Neuralgia
Acronym: CryoGem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 630286
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoneurolysis (Experimental)
  Interventions: Device: Cryoneurolysis
- Stimulation (Sham Comparator)
  Interventions: Device: Stimulation

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis
  Arms: Cryoneurolysis
Device: Stimulation — Stimulation
  Arms: Stimulation

SUMMARY:
The CryoGem Trial is a research study that tests a freezing technique called cryoneurolysis to see if it helps relieve pain in adults with trigeminal neuralgia. Trigeminal neuralgia is a condition that causes severe facial pain. In this study, we want to find out if the freezing technique is effective and safe. We will do this by comparing two groups of adults with trigeminal neuralgia. One group will receive the actual treatment, while the other group will receive a fake treatment called a sham. Neither the participants nor the assessors will know which group they are in (this is called a blinded study). For the next four weeks, participants in both groups will continue recording their headaches without knowing which treatment they are receiving. After this initial period, there will be an extension period where all participants can receive treatment as needed for up to two years. The results of this study will help us decide if the freezing technique is a viable treatment option for trigeminal neuralgia. Our main goal is to see how many people in each group have a significant reduction in pain (at least 75% less pain). We will also record other important information about the participants.

We are looking to recruit up to 24 adults with trigeminal neuralgia to take part in this study. All participants will keep a daily diary for two weeks to track their headaches before starting the treatment. Then, they will be randomly assigned to either the treatment group or the sham group.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years at the time of signing the informed consent
2. A diagnosis of primary (classic and idiopathic) trigeminal neuralgia affecting the mandibular and/or maxillary division, verified by a neurologist
3. Ability to subclassify the trigeminal neuralgia according to the The International Classification of Headache Disorders, 3rd edition, i.e. sufficient magnetic resonance (MR) evaluation is mandatory
4. History of minimum mean of three trigeminal neuralgia related pain paroxysms per day last 4 weeks
5. History of minimum average daily pain intensity NRS score (ADP) of 4 to10 last 4 weeks
6. In baseline minimum average daily pain intensity NRS score (ADP) of 4 to 10
7. In baseline minimum mean of three trigeminal neuralgia related pain paroxysms per day
8. Treatment refractory as defined in this study as failure to respond, pending an adequate trial in the opinion of the investigator, contraindications or intractable side effect to one of two medications:

   1. Carbamazepine
   2. Oxcarbazepine
9. Unaltered prophylactic TN medication regime 2 weeks prior to baseline, and be willing to keep regime unaltered during the baseline and the blinded study period.
10. Be an appropriate candidate for the study intervention required in this study on the basis of the clinical judgment of the investigator
11. Capable of giving signed informed consent as which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Diagnosed with demyelinating inflammatory disorders such as e.g. multiple sclerosis.
2. Other pain conditions, not intended to be treated in this study, that in the opinion of the investigator could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints.
3. High probability of neurological deterioration due to other medical conditions, that in the opinion of the investigator may confound outcome assessment.
4. Patients exhibiting a high degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator.
5. Other coexisting current medical conditions, including, but not limited to, bleeding diathesis and thrombophilia, that presents excess procedural risk, in the opinion of the investigator.
6. Have within 6 months of enrollment a significant untreated addiction to dependency- producing medications, alcohol, or illicit drugs.
7. Abnormal pain behavior, inappropriate medication use and/or unresolved psychiatric illness, that in the opinion of the investigator are significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome.
8. Subject has had previous radiofrequency ablation (including non-lesional pulsed radiofrequency), balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of the Gasserian ganglion.
9. Subject has had previous radiofrequency ablation (including non-lesional pulsed radiofrequency), balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of a division or branch of the trigeminal nerve being targeted in this study.
10. Facial anomaly or trauma which renders the planned procedure difficult.
11. Subject currently has an active oral or dental abscess or a local infection at the site of injection based on present symptoms.
12. Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past 6 months.
13. Current participation in another treatment study
14. Sensory deficits and/or pain configuration supporting, in the opinion of the neurologist, trigeminal neuropathy as more likely diagnosis.
15. Patients with any kind of conductive implant with contraindication for nerve stimulation according to study innervation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Average daily pain | Weeks 3 - 4 post-intervention compared to baseline
  Difference in number of treatment responders (≥ 75% reduction in the mean average daily pain intensity on a NRS score) at weeks 3 - 4 post-intervention for paroxysmal pain corresponding to the treated branch compared to baseline in the treatment versus the sham group.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 1-4
  Occurrence of treatment-emergent adverse events and serious adverse events.

SECONDARY OUTCOMES:
50% responders | Weeks 3 - 4 post-intervention compared to baseline
  Difference in number of treatment responders (≥ 50% reduction in the mean average daily pain intensity on a Numeric Rating Scale (NRS) score at weeks 3 - 4 post-intervention for paroxysmal pain corresponding to the treated branch compared to baseline) in the treatment versus the sham group.
100% responders | Weeks 3 - 4 post-intervention compared to baseline
  Difference in number of complete responders (100% reduction in the mean average daily pain intensity on a NRS score at weeks 3 - 4 post-intervention for paroxysmal pain corresponding to the treated branch compared to baseline) in the active arm versus the sham arm.
Patient Global Impression of Change (PGI-C) scale responders (a PGI- C responder is defined as having a response of "much improved" or "very much improved" at week 4.) | Week 4
  Difference in number of PGI-C responders corresponding to the treated branch at week 4 in the active arm versus sham arm.
Barrow Institute of (BNI- P) responders (a clinically significant response is defined as having BNI I - BNI IIIb at week 4). | Week 4 in the active arm versus sham arm.
  Difference in number of clinically significant BNI-P responders at week 4 in the active arm versus sham arm.
Barrow Institute of (BNI- P) excellent responders (excellent response is defined as having BNI I - BNI II at week 4). | Weeks 3 - 4 post-intervention compared to baseline
  Difference in number of excellent BNI-P responders at week 4 in the active arm versus sham arm.
Penn Facial Pain Scale- Revised (PENN-FPS-R) score. | Week 4 post-intervention compared to baseline
  Difference in reduction of PENN-FPS-R from baseline to week 4 in the active arm versus sham arm.
Change in mean average daily pain intensity NRS score (ADP) in the active versus sham arm. | Weeks 3 - 4 post-intervention compared to baseline
  Difference in reduction mean average daily pain intensity NRS score (ADP) corresponding to the treated branch at weeks 3 - 4 compared to baseline in the active arm versus the sham arm.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olavs University Hospital, Trondheim, Norway